CLINICAL TRIAL: NCT02650960
Title: Life Balance and Bimanual Activities After Stroke
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Geert Verheyden, Professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S58670
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The Flemish version of the Life Balance Inventory (LBI), measuring central constructs of life balance, will be validated in a stroke population. Upon approval by the ethical committee, stroke patients will be recruited when they are at least six months post stroke (n = 30). The LBI will be administered twice with one week interval, and demographic, socio-economic variables and other measures of health related quality of life will be collected.

Next, an observational prospective longitudinal study will be set up. We will recruit stroke patients in three rehabilitation centers within one week after admission in the rehabilitation center. Patients will undergo a baseline evaluation and will be re-assessed at discharge from the rehabilitation center, at six months and at 12 months post stroke. A standardized clinical assessment battery, measuring motor, sensory, cognitive, mental and functional outcomes as well as personal and environmental factors will be administered. This observational study will explore recovery patterns of bimanual activities after stroke from baseline evaluation to six and 12 months after stroke. Also the predictive value of motor, sensory, cognitive and mental outcomes on bimanual activities at six and 12 months post stroke is studied, based on data collected on admission to the rehabilitation center. Finally, changes over time in life balance and its determinants will be examined at six and 12 months post stroke. The predictive value of motor, cognitive and functional outcomes on life balance at one year post stroke will be examined, based on data collected on admission to the rehabilitation center. Furthermore the influence of bimanual activities on life balance will be explored in the chronic stage after stroke.

ELIGIBILITY:
Inclusion Criteria:

* first-ever stroke, as defined by the WHO criteria
* assessed and included within the first week after admission in the rehabilitation center and within the first six weeks after stroke onset
* unilateral motor impairment in the upper limb (UL - Fügl-Meyer score ≤ 60)
* minimally 18 years old
* substantial cooperation to perform the assessments
* written informed consent

Exclusion Criteria:

* other neurological impairments with permanent damage such as multiple sclerosis or Parkinson's disease
* a subdural hematoma, tumor, encephalitis or trauma that lead to similar symptoms as a stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a first-ever stroke (n=120) will be recruited consecutively by admission in three rehabilitation centers in Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Adult Assisting Hand Assessment - Stroke | 12 months post stroke
  observation based performance assessment
Life Balance Inventory | 12 months post stroke
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Principal Investigator — KU Leuven
Locations (3):
- Belgium (3):
  - RevArte, Antwerp
  - Jessa Hospitals, Herk-de-Stad
  - UZ LEuven, Leuven